CLINICAL TRIAL: NCT04040361
Title: Efficacy and Safety of Neoadjuvant Therapy of Pembrolizumab Combined With Ramucirumab for PD-L1 Positive Stage IB-IIIA Lung Cancer: An Open-label Single-arm Phase II Study
Brief Title: Neoadjuvant Therapy of Pembrolizumab + Ramucirumab for PD-L1 Positive Stage IB-IIIA Lung Cancer (EAST ENERGY)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Masahiro Tsuboi (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor-Investigator, Masahiro Tsuboi, Director of Division of Thoracic Surgery, National Cancer Center Hospital East
Organization: National Cancer Center Hospital East (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPOC1710
Record Dates: First submitted 2019-07-29; First posted 2019-07-31 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Non-small Cell Lung Cancer Stage IB; Non-small Cell Lung Cancer Stage II; Non-small Cell Lung Cancer Stage ⅢA
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Ramucirumab; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab+Ramucirumab+Surgery (Experimental): Pembrolizumab and Ramucirumab will be administered simultaneously for non small cell lung cancer patients for 2 cycles before surgery.
  Interventions: Drug: Pembrolizumab; Drug: Ramucirumab; Procedure: Surgery

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab will be administered as a dose of 200mg as a 30-minutes IV infusion, Q3W
  Other Names: MK3475
Drug: Ramucirumab — Ramucirumab will be administered as a dose of 10mg/kg as a 60-minutes IV infusion, Q3W
  Other Names: LY3009806
Procedure: Surgery — Surgery to be performed is lobectomy or more extensive lung resection and lymph node dissection

SUMMARY:
The efficacy and safety of the neoadjuvant therapy of pembrolizumab+ ramucirumab

DETAILED DESCRIPTION:
To demonstrate the antitumor activity and safety of neoadjuvant pembrolizumab plus ramucirumab followed by surgery in patients with PD-L1 positive stage IB-IIIA non-small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 20 years of age on the day of signing informed consent
2. Previously untreated and histologically proven NSCLC harboring PD-L1 expression (≥1% in a biopsy specimen), as measured by immunohistochemistry (22C3).
3. Resectable clinical stage IB-IIIA NSCLC carefully evaluated by experienced thoracic surgeons. (If N2 disease is suspected, the histological or cytological confirmation is mandatory) (UICC version 8)
4. Pulmonary resection more than lobectomy and lymph node dissection is considered to be possible for complete resection of the tumor.Be able to undergo protocol therapy, including necessary surgery.
5. Has adequate pulmonary function for pulmonary resection. Predicted postoperative FEV1.0 is 800 mL or more. ｛(predicted postoperative FEV1.0) = (preoperative FEV1.0) x (18-number of resected segment) / 18｝
6. ECOG performance status of 0 to 1.
7. Has measurable disease as defined by RECIST 1.1 as determined by investigator.
8. Has adequate organ function as defined in the following criteria. Clinical test data must meet the following criteria within 14 days of the registration. The registration day is the standard, including the same day of the week two weeks prior.

   a Neutrophil count: ≥ 1500/mm3 b Hemoglobin (Hb) ≥ 9.0 g/dL c Platelet count: ≥ 10.0 × 104/mm3 d AST (SGOT) ≤ 100 IU/L e ALT (SGPT): ≤ 100 IU/L f Total bilirubin: ≤ 1.5 mg/dL (Total bilirubin: ≤ 3.0 mg/dL for patient with Gilbert's syndrome) g Creatinine: CRE ≤ 1.5 mg/dL, or creatinine clearance of 40 mL/minute or higher [Even when the value is less than 40 mL/min in the Cockcroft-Gault equation, if the measured value from a 24-hour urine collection is 40 mL/min or higher, the patient qualifies.] * Cockcroft-Gault equation: Male: Ccr=｛(140-age) × body weight (kg)｝/｛72 × serum CRE value (mg/dL）｝Female: Ccr=0.85 × ｛(140-age) × body weight (kg)｝/｛72 × serum CRE value (mg/dL) h SpO(2) ≥ 92% (room air) i International normalized ratio (INR) ≤ 1.5 j PTT(aPTT) ≤ 1.5 × ULN k Urinary protein ≤1+ (if it is ≥2+, store the urine for 24 hours, and if the urinary protein is <1,000 mg, the patient is qualified).
9. Female who are likely to become pregnant are negative with pregnancy tests (urine or serum) within 7 days prior to enrollment. They agree to conduct proper contraception (total abstinence, intrauterine contraceptive device, hormone release system, or contraceptive implant and oral contraceptive) for both men and women during the trial and from the final investigational dosing up to 120 days
10. The participant is willing and able to provide written informed consent/assent for the trial.

Exclusion Criteria:

1. Has one of the following tumor locations/types:

   * NSCLC involving the superior sulcus
   * Large cell neuro-endocrine cancer (LCNEC)
   * Sarcomatoid tumor
   * Synchronous lung cancer (within 5 years), current non-pure GGN on TSCT, or pure GGN with 15mm or more on TSCT
2. Has an active infection requiring systemic therapy.
3. Has an active autoimmune disease that has required systemic treatment in past 2 years (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
4. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (dose exceeding 10mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of trial drug.
5. Has a known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
6. Hypersensitivity or allergy to pembrolizumab, ramucirumab, or any of their excipients.
7. Has a known history of, or any evidence of active, interstitial lung disease.
8. Has a hypertension that is difficult to control (systolic blood pressure ≥160 mmHg and diastolic blood pressure ≥90 mmHg) despite treatment with several hypotensive agents.
9. Has an acute coronary syndrome (including myocardial infarction and unstable angina), and with a history of coronary angioplasty or stent placement performed within 6 months before enrollment
10. Has a history of New York Heart Association congestive heart failure of grade II or above, unstable angina, myocardial infarction within the past 6 months, or serious cardiac arrhythmia associated with significant cardiovascular impairment within the past 6 months
11. Has a severe (hospitalization required) complications (intestinal palsy, intestinal obstruction, pulmonary fibrosis, diabetes difficult to control, heart failure, myocardial infarction, unstable angina, renal failure, liver failure, liver cirrhosis, mental disease, cerebrovascular disease etc).
12. Has a known history of human immunodeficiency virus (HIV) infection. No HIV resting is required unless mandated by local health authority.
13. Has a known history of active TB (Bacillus Tuberculosis)
14. Positivefor HBs antigens, HBs antibodies, and HBc antibodies. However, if positive for HBs and/or HBc antibodies, the patient can be registered as long as they are negative for HBV-DNA.
15. Positive for HCV antibody. However, if positive for HCV antibody, the patient can be registered as long as they are negative for HCV-RNA.
16. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
17. Has a known additional malignancy that is progressing or requires active treatment within the past (5 years) or received anti-cancer drug including hormone therapy.

    Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, bladder carcinoma, or carcinoma in situ (eg, in situ cervical cancer, breast carcinoma, CIS and AIS of the lung) that have undergone potentially curative therapy are not excluded.
18. Has received a live vaccine within 30 days prior to the first dose of trial drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist) are live attenuated vaccines and are not allowed.
19. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the screening or screening visit through 120 days after the last dose of trial treatment.
20. Has history of hemoptysis (more than 1/2 cups in teaspoon) in 2 months before registration, or invasion of major vessels by cancer or major vessel narrowing is recognized on the image.
21. Image shows cavity formation in the tumor.
22. Is considered highly likely to have complications related to bleeding.

    * Obvious tumor invasion to the chest great vessel, cavity formation of the lung lesion, or the existence of obvious thrombus on the image are recognized, etc.
23. Has past history of gastrointestinal perforation, peptic ulcer, diverticulosis or fistula within 6 months.

    ※ As for peptic ulcer, registration is permitted when disease condition is controlled by appropriate treatment.
24. Has a history of pulmonary embolism / deep vein thrombosis, or other thromboembolism within 3 months before registration.
25. Received major surgery within 28 days before registration, or received procedures for placement of subcutaneous venous access devices within seven days before registration.
26. Severe wounds, ulcers or fractures within 28 days before registration.
27. Has undergone long-term treatment using aspirin, nonsteroidal anti-inflammatory drugs (such as ibuprofen, naproxen), dipyridamole, clopidogrel or similar drugs. However, use of aspirin up to 325 mg / day once a day is acceptable.
28. Patients who are receiving anticoagulant therapy and whose dose of oral anticoagulant or low molecular weight heparin is not stable. In case of taking warfarin, registration is permitted if there is no active bleeding or no risk of bleeding.
29. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of registration.

    Note: Participants who have entered the follow-up phase of an investigational trial may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
30. Has no intention to comply with the study protocol or it is impossible to comply.
31. Investigator or clinical trial doctor judged unsuitable as subject of this trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-11-30 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Major pathologic response (MPR) rate by central review | 1 year 7 months
  Determination of major pathologic response rate is based on the method by Hellmann et al. on the pathological section. The percentage of residual tumor cells is calculated as viable tumor cells / tumor area × 100 (%). Tumor area includes viable tumor cells and interstitial tissue such as fibrosis, necrosis, and inflammatory cells.

SECONDARY OUTCOMES:
Proportion of incidence of adverse events | 1 year 7 months
  The incidences and types of adverse events that occur during neoadjuvant therapy and perioperative period (within postoperative 30 days and 90 days) will be evaluated according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Major pathological response (MPR) rate by institutional report | 1 year 7 months
  Determination of major pathologic response rate by institutional report
Pathological complete response rate (pCR rate) | 1 year 7 months
  Pathological complete response rate (pCR rate)
Pathological complete resection rate (R0 rate) | 1 year 7 months
  Pathological complete resection rate (R0 rate)
Objective response rate (ORR) according to RECIST and iRECIST | 1 year 7 months
  Objective response rate (ORR) according to RECIST and iRECIST
Overall survival (OS) | 5 years
  Overall survival (OS)
Recurrence-free survival (RFS) | 5 years
  Recurrence-free survival (RFS)

CONTACTS AND LOCATIONS:
Overall Officials: Masahiro Tsuboi, Dr, Principal Investigator — National Cancer Center Hospital East
Locations (2):
- Japan (2):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Tokyo Medical University Hospita, Shinjuku-Ku, Tokyo